CLINICAL TRIAL: NCT05120999
Title: Comparison of Onset of Neuromuscular Blockade With Electromyographic and Acceleromyographic Monitoring: A Prospective, Randomized Trial
Brief Title: Comparison of Onset of Neuromuscular Blockade With Electromyographic and Acceleromyographic Monitoring
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 21-007425
Record Dates: First submitted 2021-10-26; First posted 2021-11-16 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Neuromuscular Blockade
Keywords: neuromuscular blockade

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dominant hand: Application of either TetraGraph or TOFScan device on dominant hand
  Interventions: Device: Train of four measurement
- Non-Dominant hand: Application of either TetraGraph or TOFScan device on non-dominant hand
  Interventions: Device: Train of four measurement

INTERVENTIONS:
Device: Train of four measurement — Use of either TetraGraph or TOFScan to measure the neuromuscular blockade

SUMMARY:
The purpose of this research is to use 2 devices to compare the difference in the amount of time it takes for each device to register complete muscle relaxation after the muscle relaxing medication is given. The comparison will be made by using electromyographic (EMG), such as TetraGraph, and acceloromyographic (AMG), such as TOFScan, monitors at the time of insertion of breathing tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate and provide an informed consent.
* Patients undergoing elective surgical procedures that require use of NMBA agents (rocuronium) administered intraoperatively.

Exclusion Criteria:

* Patients with disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
* Patients with systemic neuromuscular diseases such as myasthenia gravis.
* Patients with significant organ dysfunction that can significantly affect pharmacokinetics of neuromuscular blocking and reversal agents; i.e., severe renal impairment or end-stage liver disease.
* Patients having surgery that would involve prepping the arm into the sterile field.
* Patients receiving a rapid sequence induction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Qualified participants will be invited to participate in this study regardless of gender, sex, race, or religion.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Time difference | During the initiation of anesthesia period
  Compare time difference from neuromuscular blockade agent administration to neuromuscular blockade onset

SECONDARY OUTCOMES:
Intubating conditions | During the initiation of anesthesia period
  Assess intubating conditions once a complete neuromuscular blockade has been achieved either by TetraGraph or TOFScan measurements

CONTACTS AND LOCATIONS:
Overall Officials: J. Ross Renew, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Chaves-Cardona HE, Fouda EA, Hernandez-Torres V, Torp KD, Logvinov II, Heckman MG, Renew JR. Comparison of onset of neuromuscular blockade with electromyographic and acceleromyographic monitoring: a prospective clinical trial. Braz J Anesthesiol. 2023 Jul-Aug;73(4):393-400. doi: 10.1016/j.bjane.2023.04.004. Epub 2023 May 1. PMID 37137388
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials